CLINICAL TRIAL: NCT00552630
Title: A Phase 2/3 Trial of d-Penicillamine Chelation in Lead-Poisoned Children
Brief Title: Penicillamine Chelation for Children With Lead Poisoning
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Bezoloven, Inc. (Industry)
Responsible Party: Michael Shannon, MD, Children's Hospital Boston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3361; 1R01FD003361-01A1 (FDA)
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2007-12

CONDITIONS: Lead Poisoning; Vitamin D Deficiency
Keywords: lead poisoning; chelation
MeSH Terms: conditions — Lead Poisoning; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): This group will receive d-penicillamine for 6 weeks
  Interventions: Device: d-penicillamine
- 2 (Placebo Comparator): This group will receive placebo for 6 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Device: d-penicillamine — d-penicillamine twice daily, 15 mg/kg/day, for 6 weeks
  Arms: 1
Drug: placebo — placebo with same characteristics as drug
  Arms: 2

SUMMARY:
Childhood Lead Poisoning is a widespread disease that has few effective treatments. The specific aims of this proposed clinical trial are threefold:

* To determine whether a six-week course of a newly formulated d-penicillamine suspension will effectively reduce blood lead level in children aged 6 months to 16 years with blood lead levels of 15-25 μg/dL.
* To determine whether d-penicillamine chelation produces a sustained reduction in blood lead level in comparison with succimer and other lead chelators which always produce a significant post-treatment "rebound".
* To determine whether chelation with d-penicillamine improves the physiologic disturbances that can be measured in children with blood lead levels in this range.

DETAILED DESCRIPTION:
Approximately 300,000 children in the US have elevated blood lead levels (10 mcg/dl or greater). Lead poisoning in children is unequivocally harmful, producing the neurodevelopmental consequences of cognitive losses, attentional difficulties and behavioral disturbances, including antisocial or delinquent tendencies. Non-neurodevelopmental consequences of lead poisoning include impairment of heme synthesis, reduction in 1- hydroxylation of 25(OH) - cholecalciferol (the Vitamin D precursor) and renal injury that results in microproteniuria, an increased risk of hypertension and a greater likelihood of renal failure in adulthood. Despite these well-defined toxicities, treatments for childhood lead poisoning have been inadequate. Currently, chelation therapy is uniformly recommended only for children with severe lead poisoning (blood lead > 45 mcg/dl). Approved chelating agents for severe plumbism are CaNa2EDTA and succimer. For children with blood lead levels less than 45 mcg/dl treatment is fraught with difficulties including inconsistent recommendations by clinical experts, lack of proven benefit of chelation and the absence of a chelating agent approved for use in this range. d-Penicillamine is a lead chelator that has been used off-label for almost 4 decades. Several studies have suggested that d-penicillamine is both safe and effective in the treatment of low-level lead poisoning. We propose to evaluate, in a Phase II/III randomized, placebo-controlled clinical trial, the effectiveness of d-penicillamine in 50 children aged 6 months to 16 years with blood lead levels 15-25 mcg/dl. The d-penicillamine product will be a newly developed, IND-approved liquid formulation. The study will be performed in the Pediatric Environmental Health Center of Children's Hospital Boston. The primary outcome measure will be the ability of a 6-week course of d-penicillamine to produce sustained reductions in blood lead level. Secondary outcome measures will be normalization of non-neurodevelopmental physiologic aberrations known to occur with lead poisoning, specifically abnormalities in heme and Vitamin D synthesis. If this clinical trial demonstrates safety and efficacy, d-penicillamine will potentially provide another option among the limited treatment choices for lead-poisoned children. This trial will also provide a basis for examining the drug's efficacy in improving neurodevelopment outcome in children exposed to harmful amounts of lead.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects will be children 6 months to 16 years of age with blood lead level 15-25 mcg/dL on two separate occasions separated by at least two weeks

Exclusion Criteria:

* allergic to d-penicillamine
* renal insufficiency
* taking immunosuppressive agents
* pre-existing idiopathic thrombocytopenia (platelet count < 100,000/mm3) or leukopenia (WBC count < 5,000/mm3 or polymorphonuclear leukocyte count < 1000/mm3)
* blood lead level on the day of the initial clinic visit is below15 μg/dL or above 25 μg/dL
* blood lead level at the two-week follow up visit rises above 25 mcg/dL or falls below 15 mcg/dL
* currently undergoing chelation or have had chelation therapy in the previous two months

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-09

PRIMARY OUTCOMES:
• To determine whether a six-week course of a newly formulated d-penicillamine suspension will effectively reduce blood lead level in children aged 6 months to 16 years with blood lead levels of 15-25 μg/dL. | 6 weeks

SECONDARY OUTCOMES:
To determine whether d-penicillamine produces a sustained reduction in blood lead level and improves the physiologic disturbances that can be measured in children with blood lead levels in this range. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Shannon, MD, Study Director — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States